CLINICAL TRIAL: NCT02204436
Title: Clinical Study for the Evaluation of the Depigmenting Activity of a Cosmetic Product on Spotted Hand Skin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Derming SRL (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E3013
Record Dates: First submitted 2014-07-18; First posted 2014-07-30 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-03

CONDITIONS: Healthy
Keywords: hyperpigmentation; depigmenting treatment; hand
MeSH Terms: conditions — Hyperpigmentation | interventions — Emulsions; Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Emulsion and gel (Other): A fixed similar quantity of both emulsion and gel were applied consequentially on the hand twice a day, in the morning and in the evening (preferentially always at the same hour), with a mild massage, until complete absorption, for 8 weeks.
  Interventions: Other: Emulsion and gel

INTERVENTIONS:
Other: Emulsion and gel — A fixed similar quantity of both emulsion and gel were applied consequentially on the hand twice a day, in the morning and in the evening (preferentially always at the same hour), with a mild massage, until complete absorption, for 8 weeks.

SUMMARY:
Aim of the study was to evaluate by instrumental measurements the depigmenting activity of a cosmetic treatment for spotted hand skin; in particular it was investigated the synergic activity of an emulsion, with clarifying-antioxidant activity combined with an activator gel, with hydration and keratolytic activity.

Female healthy volunteers aged 45-65 years old, presenting senile lentigo on the hands, were included in the study.

It was also aim of this study to evaluate treatment efficacy and cosmetic acceptability by the volunteers and tolerance both by investigator and volunteers.

DETAILED DESCRIPTION:
The following instrumental evaluations were performed in basal conditions (T0 - before product use), after 4 (T4) and 8 week-treatment (T8):

* Image analysis with UV flash (Wood's light)
* Photographic recovery
* Skin spots image analysis
* Skin colour evaluation
* Spectrophotometry (skin brightness)
* Optical colorimetry (spots colour)

At the end of the study (T8), each volunteer filled a questionnaire regarding:

* the efficacy of the study product (skin brightness and hydration, spots dimensions and colour intensity - score: very marked; marked; medium; light; absent)
* the cosmetic acceptability of the study product: colour and perfume before and after application, consistency, spreadability, absorption, effect on the skin, greasiness and presence of product residues (score: negative; medium; good; excellent) the product tolerance (score: bad; poor; medium; good; excellent).

At the end of the study the investigator assessed the treatment tolerance considering the possible appearance of related adverse events as bad, poor, medium, good, excellent.

ELIGIBILITY:
Inclusion Criteria:

* female healthy subjects
* age 45-65 years
* presence of moderate senile lentigo on the back of the hands
* accepting to not receive any drugs/cosmetic/chemical or physical treatment (peeling, intradermal implants etc.) able to change the skin characteristics during the entire duration of the study
* accepting to use the study product according to the instruction received by the investigator
* accepting not to expose to strong UV irradiation (UV session, or sun bathes) during the entire duration of the study
* subject agreeing not to use anti-spots products/treatments during the month preceding the test
* accepting to sign the Informed Consent Form

Exclusion Criteria:

* pregnancy
* lactation
* sensitivity to the test product or its ingredients
* subjects whose insufficient adhesion to the study protocol is foreseeable
* participation in a similar study actually or during the previous 3 months
* dermatological disease (dermatitis; presence of cutaneous disease on the tested area, as lesions, scars, malformations)
* clinical and significant skin condition on the test area (e.g. active eczema, dermatitis, psoriasis. etc.)
* diabetes
* endocrine disease
* hepatic disorder
* renal disorder
* cardiac disorder
* pulmonary disease
* cancer
* neurological or psychological disease
* inflammatory/immunosuppressive disease
* drug allergy
* systemic corticosteroids
* aspirin or non-steroid anti-inflammatory drugs (FANS)
* anti-histaminic, narcotic, antidepressant, immunosuppressive drugs (with except of contraceptive or hormonal treatment starting from at least 1 year)
* assumption of drugs able to influence the test results in the investigator opinion

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Skin spots image analysis: change from baseline (T2, T4 and T8 vs. T0) | after 2, 4 and 8-week-treatment
  Skin spots area was measured on the pre-selected images performed with or without Wood's lamp. The measure of skin spots area was performed by means of an image analysis software, with a function called "magic wand". Based on the colour similarities or on the difference of intensity ranges between the selected pixels (with a specified tolerance interval) the magic wand automatically traced the outline of the spot and measured the selected area (pixel2).

SECONDARY OUTCOMES:
Spectrophotometric evaluation: change from baseline (T2, T4 and T8 vs. T0) | after 2, 4 and 8-week-treatment
  Skin brightness was measured by a visible-UV-IR (λ from 300 to 900 nm) spectrophotometer which uses a tungsten halogen lamp and a deuterium lamp in accordance with CIE (Commission Internationale de l'Eclarage), the main international organisation concerned with colour and colour measurement. Lamps were switched on 30 minutes before instrument use in order to join a stable emission. Measurement angle was 90° (position of the probe on the skin) and measured area was 2 mm2; used wavelength range was 380-780 nm corresponds to the visible light spectrum.
Optical colorimetry: change from baseline (T2, T4 and T8 vs. T0) | after 2, 4 and 8 week-treatment
  Measurement of spots colour were performed by a tri-stimulus colorimeter equipped with three special filters to obtain R,G,B values in accordance with CIE (Commission Internationale de l'Eclarage), the main international organisation concerned with colour and colour measurement. CIE L*a*b* system (CIELAB) is the most complete colour-space specified by the CIE (1976). It describes all the colours visible to the human eye; the three coordinates of L*a*b* represent the lightness of the colour (L* = 0 yields black and L* = 100 indicates diffuse white; specular white may be higher), its position between red/magenta and green (a*, negative values indicate green while positive values indicate magenta) and its position between yellow and blue (b*, negative values indicate blue and positive values indicate yellow).

CONTACTS AND LOCATIONS:
Overall Officials: Adele Sparavigna, Doctor, Principal Investigator — Derming SRL
Locations (1):
- DermIng SRL, Monza, Monza, Italy

REFERENCES:
- [Background] Asawanonda P, Taylor CR. Wood's light in dermatology. Int J Dermatol. 1999 Nov;38(11):801-7. doi: 10.1046/j.1365-4362.1999.00794.x. No abstract available. PMID 10583611
- [Background] Asserin J., Heusèle C., André P. , Preece S., Schnebert S. , Taieb A. Comparison of two techniques used in the evaluation of the depigmentation effect of cosmetic products on brown spots, 2004
- [Background] Claridge E, Cotton S, Hall P, Moncrieff M. From colour to tissue histology: Physics-based interpretation of images of pigmented skin lesions. Med Image Anal. 2003 Dec;7(4):489-502. doi: 10.1016/s1361-8415(03)00033-1. PMID 14561553
- [Background] Claridge E, Preece SJ. An inverse method for the recovery of tissue parameters from colour images. Inf Process Med Imaging. 2003 Jul;18:306-17. doi: 10.1007/978-3-540-45087-0_26. PMID 15344467
- [Background] Curry AS, Gettings SD, McEwen GN CTFA safety testing guidelines. The Cosmetic, Toiletry and Fragrance Association, Washington, 1991
- [Background] Fernay, Voltaire The World Medical Association (1989) "World Medical Association Declaration of Helsinki", Hong-Kong
- [Background] Fullerton A, Fischer T, Lahti A, Wilhelm KP, Takiwaki H, Serup J. Guidelines for measurement of skin colour and erythema. A report from the Standardization Group of the European Society of Contact Dermatitis. Contact Dermatitis. 1996 Jul;35(1):1-10. doi: 10.1111/j.1600-0536.1996.tb02258.x. PMID 8896947
- [Background] Gilchrest BA, Fitzpatrick TB, Anderson RR, Parrish JA. Localization of malanin pigmentation in the skin with Wood's lamp. Br J Dermatol. 1977 Mar;96(3):245-8. doi: 10.1111/j.1365-2133.1977.tb06132.x. PMID 857837
- [Background] Gupta LK, Singhi MK. Wood's lamp. Indian J Dermatol Venereol Leprol. 2004 Mar-Apr;70(2):131-5. No abstract available. PMID 17642589
- [Background] Matts Paul J., Carey Jeremy, Cotton Symon D. Chromophore Mapping: a New Technique to Characterize Aging Human Skin, In Vivo. American Academy of Dermatology 2005
- [Background] Matts PJ, Dykes PJ, Marks R. The distribution of melanin in skin determined in vivo. Br J Dermatol. 2007 Apr;156(4):620-8. doi: 10.1111/j.1365-2133.2006.07706.x. PMID 17493065
- [Background] Moncrieff M, Cotton S, Claridge E, Hall P. Spectrophotometric intracutaneous analysis: a new technique for imaging pigmented skin lesions. Br J Dermatol. 2002 Mar;146(3):448-57. doi: 10.1046/j.1365-2133.2002.04569.x. PMID 11952545
- [Background] Rieger M.M., Battista G.W. Some experiences in the safety testing of cosmetics J. Soc. Cosmet. Chem. 15:161 -172 , 1964
- [Background] Rigano L. "Evaluation of the efficacy of a whitening product" ISPE Institute of Skin and Product Evaluation - March 15th 2007
- [Background] Sachs L. Applied statistics: a handbook of techniques Heidelberg: Springer, 1981:536-539
- [Background] Taelman M-C, Dederen J. C. Relative performance testing of formulations: emulsifiers Cosmetics &Toiletries magazine August 2000; 115: 37-42
- [Background] Takiwaki H. Measurement of skin color: practical application and theoretical considerations. J Med Invest. 1998 Feb;44(3-4):121-6. PMID 9597799
- [Background] Zonios G, Bykowski J, Kollias N. Skin melanin, hemoglobin, and light scattering properties can be quantitatively assessed in vivo using diffuse reflectance spectroscopy. J Invest Dermatol. 2001 Dec;117(6):1452-7. doi: 10.1046/j.0022-202x.2001.01577.x. PMID 11886508
- See also: Investigator center — http://www.derming.com
- See also: Sponsor — http://www.giulianipharma.com/